CLINICAL TRIAL: NCT06720610
Title: Comparison of the Effectiveness of Vonoprazan and Esomeprazole in Improving Initial Symptoms in Patients with Erosive Esophagitis: a Double-Blind Randomized Trial
Brief Title: Indonesian Study of Vonoprazan Vs Esomeprazole in Erosive Esophagitis
Acronym: INVEST
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ari Fahrial Syam, Dean of Faculty of Medicine Universitas Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INVEST01; 24-08-1382 (Other: The Ethics Commitee of the Faculty of Medicine, University of Indonesia - Cipto Mangunkusumo Hospital)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Erosive Esophagitis
Keywords: erosive esophagitis; vonoprazan; esomeprazole; gerd-q
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vonoprazan (Experimental): Each randomized patients will consume 20mg of vonoprazan once a day for 14 days consecutively
  Interventions: Drug: Vonoprazan 20 mg
- Esomeprazole (Active Comparator): Each randomized patients will consume 40mg of esomeprazole once a day for 14 days consecutively
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Vonoprazan 20 mg — Vonoprazan PO, 20mg, once a day, 14 days.
  Other Names: vocinti
  Arms: Vonoprazan
Drug: Esomeprazole — Esomeprazole PO, 40mg, once a day, 14 days
  Other Names: Esomeprazole generic
  Arms: Esomeprazole

SUMMARY:
The goal of this clinical trial is to compare drug vonoprazan vs esomeprazole effectiveness to relieve early symptoms in Erosive Esophagitis Patients. It will also learn about the safety of both modalities. The main questions it aims to answer are:

How does the effectiveness of Vonoprazan compare with Esomeprazole in improving early symptoms of erosive esophagitis patients in the Indonesian population?

Researchers will compare drug vonoprazan to a esomeprazole with a look-alike packaging to see their effect to reduce early symptoms of erosive esophagitis.

Participants will:

* Take drug vonoprazan 20mg or esomeprazole 40mg one time every day for 2 weeks
* Visit the clinic once every weeks for followup (Gastro Esophageal Reflux Disease-Quetionnaire measurement)
* Keep a diary of their adverse effect occurence and every variable data based on Gastro Esophageal Reflux Disease-Questionnaire.

DETAILED DESCRIPTION:
Based on the calculation using the formula for comparing two population proportions, the minimum estimated sample size is 97 samples for each group. Considering a potential 10% drop-out rate, the estimated sample size increases to 108 samples per group. Therefore, the total minimum sample required for this study is 216 samples for both groups.

All the patients will screened using the Gastro Esophageal Reflux Disease-Quetionnaire (6 questions, 4 answer options, covering the last 7 days) and collected through RedCap. After that all eligible patients will undergo endoscopic examination that performed by gastroenterology specialists or trained internists.

Included patients who consume any Proton Pump Inhibiotr or Potassium-competitive acid blockers within 2 weeks prior to this study will undergo wash-out period for 2 weeks. Patients are monitored weekly during the wash-out period. Medication reminders are sent via instant messaging at least twice per week. Adverse Event will be monitored by research assistants in coordination with the patient's primary physician.

All the data will analyzed blindly with Chi-square or Fisher's exact test for categorical data and logistic regression for confounding factors. At the end of the study, the pharmacy team will reveal the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years with a GERD-Q score of 8.
* Diagnosed with erosive esophagitis by endoscopy. (Los Angeles Classification A-D)
* Patients are willing to undergo a series of therapeutic management.

Exclusion Criteria:

* Patients with a history of allergy to PCAB or PPI groups.
* Patients with gastric and/or duodenal ulcers.
* Patients with Helicobacter pylori infection.
* Patients with a history of significant systemic disease disorders affecting the esophagus and stomach.
* Patients with a history of malignant disease related to the esophagus and/or stomach.
* Patients with a history of esophageal and/or gastric surgery.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Symptoms Resolution of Erosive Esophagitis | 14 days (two weeks)
  Participants achieved a,
  * complete resolution if they scored a GERD-Q questionnaire of 0 from scale 0-18. - sufficient relief if they scored GERD-Q of 1 or 0 (No. 1,2,5,6)
  * persistent response if they score GERD-Q of 2 or more in any single question.

SECONDARY OUTCOMES:
Number of Participants with Adverse Event | 14 days (two weeks)
  Yes: nasopharyngitis, diarrhea, acute upper respiratory infection, lower back pain, constipation No: none of any

OTHER OUTCOMES:
Rate of Drug Compliance | 14 days (two weeks)
  Compliant (14 drugs finished in 14 days) Lack of compliance (14 drugs finished in >14 days) Non-compliant (not taking drugs)

CONTACTS AND LOCATIONS:
Overall Officials: Ari F Syam, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (5):
- Indonesia (5):
  - Hermina Jatinegara Hospital, East Jakarta, DKI Jakarta
  - Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta
  - Hermina Kemayoran Hospital, Jakarta Pusat, DKI Jakarta
  - Hermina Bekasi Hospital, Bekasi, West Java
  - Hermina Depok Hospital, Depok, West Java

IPD SHARING:
Plan to Share IPD: No